CLINICAL TRIAL: NCT00982189
Title: Cardiovascular Disease Risk Reduction for Persons With HIV Infection: a Polypill Pilot Study
Brief Title: Cardiovascular Prevention for Persons With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PCC-003
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection; Cardiovascular Disease Risk
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Pravastatin; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lisinopril (Experimental): Lisinopril 10mg once daily
  Interventions: Drug: Lisinopril
- Lisinopril Placebo (Placebo Comparator): Placebo pill (matched to lisinopril) once daily
  Interventions: Drug: Lisinopril
- Pravastatin (Experimental): Pravastatin 20mg once daily
  Interventions: Drug: Pravastatin
- Pravastatin placebo (Placebo Comparator): Placebo pill (matched to pravastatin) once daily
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Participants randomized to take pravastatin (active) or matching placebo pill once daily
  Arms: Pravastatin; Pravastatin placebo
Drug: Lisinopril — Participants randomized to take lisinopril (active) or matching placebo pill once daily
  Arms: Lisinopril; Lisinopril Placebo

SUMMARY:
This study is funded by the American Heart Association. The goal of this research is to prevent early cardiovascular damage before symptoms develop for persons with HIV infection. Evidence suggests that taking low doses of blood pressure and cholesterol medication reduces risk for heart disease in persons who are at increased risk (such as the case with HIV infection).

Participants who are taking HIV treatment with an 'undetectable' viral load, and who do NOT need treatment for high blood pressure or cholesterol may be eligible to enroll. Participants will take a low dose cholesterol medication (or placebo) and a low dose of a blood pressure medication (or a placebo), and will be seen at 3 study visits over 4 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection with viral load 'undetectable' while taking antiretroviral therapy
* Age ≥40
* Framingham risk score (FRS) ≥5%, or ≥3% with ≥5 years of exposure to antiretroviral therapy

Exclusion Criteria:

* Known cardiovascular disease or Framingham risk score (FRS) ≥20%
* Blood pressure ≥140/90
* LDL cholesterol ≥160 (with FRS <10%), or ≥130 (with FRS 10-20%)
* Currently taking, or has a medication contraindication to take, a 'statin', an ACE inhibitor, or an angiotensin receptor blocker medication
* Cirrhosis or plasma ALT/AST levels >2x upper limit of normal
* Chronic kidney disease and a creatinine >2.0mg/dL
* Triglycerides >500mg/dL

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Baker, MD, Principal Investigator — Hennepin Faculty Associates
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Baker JV, Huppler Hullsiek K, Prosser R, Duprez D, Grimm R, Tracy RP, Rhame F, Henry K, Neaton JD. Angiotensin converting enzyme inhibitor and HMG-CoA reductase inhibitor as adjunct treatment for persons with HIV infection: a feasibility randomized trial. PLoS One. 2012;7(10):e46894. doi: 10.1371/journal.pone.0046894. Epub 2012 Oct 17. PMID 23082133

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril/P-placebo: Lisinopril 10mg and placebo (matched to pravastatin) once daily
- L-placebo/Pravastatin: Placebo pill (matched to lisinopril) and Pravastatin 20mg once daily
- Lisinopril/Pravastatin: Lisinopril 10mg and Pravastatin 20mg once daily
- L-placebo/P-placebo: Placebo pill (matched to pravastatin) and placebo pill (matched to lisinopril) once daily
Period: Overall Study
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo
Started | 10 | 9 | 9 | 9
Completed | 10 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo | Total
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 9 | 9 | 37
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 47 (12) | 48 (4) | 45 (7) | 48 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1
  Male | 10 | 8 | 9 | 9 | 36
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 9 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Stated (by Self-report) That They Had Side Effects
Description: Participants were asked at each visit if they had any side effects to study medication. They provided a yes or no answer, and if yes they specified what the side effect was.
Time Frame: 4 months
Population: Number of participants who stated (by self-report) that they had side effects
Measure: Number; unit: participants
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9
participants | 1 | 0 | 2 | 1

2. Primary Outcome: Number of Participants Who Took >90% of Their Doses (by Pill Count)
Description: The number of pills missing from study medication bottles was counted by study nurses at the completion of the study. The proportion of pills taken divided by the number of days the participant was enrolled in the study was calculated, and multiplied by 100, to generate the '% of doses taken'
Time Frame: 4 months
Population: Number of participants who took >90% of their doses (by pill count)were studied. All participants who returned unused medications at end of the study were included for these analyses
Measure: Number; unit: participants
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo
Number analyzed (Participants) | 4 | 7 | 8 | 6
participants | 2 | 7 | 5 | 6

3. Primary Outcome: Change From Baseline to Month 4 in the Framingham Risk Score (FRS)
Description: The Framingham Risk Score is calculated by a published algorithm that predicts a patients risk of having a coronary heart disease event in the next 10 years. The measures that are considering in predicting this risk are: age, blood pressure, cholesterol (both total cholesterol and high-density lipoprotein cholesterol), smoking status, and use of medication to treat hypertension. This risk score can be estimated using an online calculator (http://hp2010.nhlbihin.net/atpiii/calculator.asp)
Time Frame: Change from baseline to 4 months
Population: All participants had Framingham risk score (FRS) estimated at baseline and month 4. The change from baseline to month 4 was calculated as the outcome.
Measure: Median (Inter-Quartile Range); unit: Percent probability of CHD event in 10yr
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo
Number analyzed (Participants) | 10 | 9 | 9 | 9
Percent probability of CHD event in 10yr | -1.6 [-2.3 to 1.1] | -0.7 [-2.6 to 0.4] | -1.5 [-2.1 to 0.5] | -0.3 [-0.7 to 0.2]

4. Secondary Outcome: Changes in Blood Pressure
Description: Blood pressure was assessed by standard clinical methods (i.e., the same way it is measured during a routine clinic visit)
Time Frame: change from baseline to 4 months
Population: n=17 Lisinopril vs. n=17 L-placebo The outcome is analyzed as the 'main effect' for lisinopril versus placebo, as standard for factorial study designs. Since lisinopril, but not pravastatin, influences blood pressure, the analysis defines Lisinopril and L-placebo groups by pooling across pravastatin groups (i.e., P-placebo + Pravastatin groups).
Measure: Mean (95% Confidence Interval); unit: (mmHG)
Groups:
- Lisinopril/L-placebo Treatment Effect: Lisinopril vs. Lisinopril-placebo (regardless of Pravastatin status)
Arm/Group | Lisinopril/L-placebo Treatment Effect
Number analyzed (Participants) | 34
(mmHG)
  Systolic BP | -1.8 [-9.4 to 5.8]
  Diastolic BP | -3.3 [-7.3 to 0.7]

5. Secondary Outcome: Changes in Blood Lipids
Description: Blood lipids include routine cholesterol measurements that are monitored in clinical practice. They are measured in blood after a blood draw is performed. The specific measurements include: a) total cholesterol, b) low-density lipoprotein cholesterol, c) high-density lipoprotein cholesterol, and d) triglycerides
Time Frame: change from baseline to 4 months
Population: n = 18 Pravastatin vs. n = 16 P-placebo The outcome is analyzed as the 'main effect' for pravastatin versus placebo, as standard for factorial study designs. Since pravastatin, but not lisinopril, influences cholesterol, the analysis defines Pravastatin and P-placebo groups by pooling across lisinopril groups (i.e., L-placebo + Lisinopril group).
Measure: Mean (95% Confidence Interval); unit: (mg/dL)
Groups:
- Pravastatin/P-placebo Treatment Effect: Pravastatin vs. Pravastatin-placebo (regardless of Lisinopril status)
Arm/Group | Pravastatin/P-placebo Treatment Effect
Number analyzed (Participants) | 34
(mg/dL)
  Total Cholesterol | -1.75 [-18.74 to 15.25]
  LDL-C | -0.62 [-13.22 to 11.98]
  HDL-C | 0.97 [-8.42 to 10.36]

6. Secondary Outcome: Changes in Small Artery Elasticity
Description: Small artery elasticity is a measure of vascular function, estimated through analysis of the blood pressure waveform. A sensor is placed on wrist over the radial pulse. The blood pressure waveform of the pulse is recorded and analyzed the elasticity, or compliance, of the small (and large) vasculature. Impaired artery elasticity, or increased stiffness, is an early sign of vascular disease that predicts risk for future cardiovascular events.
Time Frame: change from baseline to 4 months
Population: Analysis presents the baseline-to-month4 difference between Lisinopril versus L-placebo groups; n=17 Lisinopril vs. n=17 L-placebo Our hypothesis for this secondary outcome was the 'main effect' for Lisinopril versus placebo would reduce inflammation. There was no interaction, so analyses define Lisinopril and L-placebo groups as for outcome #4
Measure: Mean (Standard Error); unit: mL/mmHgx100
Arm/Group | Lisinopril/L-placebo Treatment Effect
Number analyzed (Participants) | 34
mL/mmHgx100 | 0.02 (0.75)

7. Secondary Outcome: Changes hsCRP (C-reactive Protein)
Description: This biomarker represents systemic inflammation within in the body.
Time Frame: change from baseline to 4 months
Population: as for outcome 6
Measure: Geometric Mean (Standard Error); unit: mcg/mL
Arm/Group | Lisinopril/L-placebo Treatment Effect
Number analyzed (Participants) | 34
mcg/mL | -1.00 (0.40)

8. Secondary Outcome: Changes IL-6 (Interleukin-6)
Description: This biomarker represents systemic inflammation within in the body.
Time Frame: change from baseline to 4 months
Population: as for outcome 6
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Lisinopril/L-placebo Treatment Effect
Number analyzed (Participants) | 34
pg/mL | -0.33 (0.24)

9. Secondary Outcome: Changes TNFa (Tumor Necrosis Factor Alpha)
Description: This biomarker represents systemic inflammation within in the body.
Time Frame: change from baseline to 4 months
Population: as for outcome 6
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Lisinopril/L-placebo Treatment Effect
Number analyzed (Participants) | 34
pg/mL | -0.14 (0.10)

ADVERSE EVENTS:
Arm/Group | Lisinopril/P-placebo | L-placebo/Pravastatin | Lisinopril/Pravastatin | L-placebo/P-placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Study was small with limited power to detect differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No